CLINICAL TRIAL: NCT03196323
Title: Development of a Behavioral Outcome Measure for Rett Syndrome (RettBe)
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: RTT5214
Record Dates: First submitted 2017-06-02; First posted 2017-06-22 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initial Cohort: In Aim 1, the investigators will evaluate psychometrically RettBe 1.0 following, in part, previous studies including our examination of anxiety instruments and adaptation of the Anxiety, Depression and Mood Scale (ADAMS) for RTT, and their adaptations of the Aberrant Behavior Checklist-Community (ABC-C) for fragile X syndrome and Down syndrome. In Aim 1, the investigators will also refine RettBe 1.0 by adding new "missing" items based on parental input or clinician (PIs of sites involved) feedback. The resulting instrument, RettBe 2.0 will be tested in Aim 2.
- Validation Cohort: Testing of RettBe 2.0 will be carried out with a new (naïve) validation cohort of 300 subjects and two raters (preferentially both parents/caregivers, alternatively one teacher or therapist), to determine inter-rater reliability. One rater, preferentially a parent, will be asked to also complete three other behavioral measures (RSBQ, ADAMS, ABC-C) for comparisons. Scores for RettBe 2.0 will be analyzed in terms of psychometric properties, as performed for RettBe 1.0. However, in addition to structure (construct validity) and content validity, the investigators will also examine convergent and discriminant validity by correlating domain RettBe 2.0 scores with those of comparable and non-comparable domain scores of the RSBQ, ADAMS, and ABC-C, respectively.

SUMMARY:
The overall purpose of this study is to develop a broad-based (i.e., multiple domains) behavioral outcome measure for children between the ages of 3-18 years with Rett syndrome (RTT). The innovative approach of this proposal consists of integrating the process of developing a behavioral questionnaire to an ongoing large-scale data collection project. The Natural History Study of Rett Syndrome and Related Disorders (RTT5211) is a project that collects data on diverse aspects of the clinical evolution of individuals with RTT and related disorders. This project will serve as the basis for recruitment of subjects and it will also provide key demographic and clinical data for cohort characterization and for determining clinical relevance of the instrument (RettBe). An initial 100-subject cohort will allow for the testing with one rater of RettBe 1.0, a 50-item questionnaire formed from existing measures, a panel of clinicians and behavioral experts in RTT, and a focus group of parents and caregivers of children with RTT. Scores on RettBe 1.0 will be statistically analyzed to determine their psychometric properties, including its content validity. Items that do not meet psychometric standards (e.g., ceiling effect) will be eliminated.

Additional items will be added if the parental survey attached to RettBe 1.0 or clinician input suggests so. The resulting modified assessment, called RettBe 2.0, will be administered to a larger (validation) cohort of 300 participants. RettBe 2.0 will also be subjected to analysis of psychometric properties. RettBe 2.0 will also be administered to two raters per subject, in order to determine inter-rater reliability. In addition, these raters will be completing other behavioral and clinical measures for further evaluating the validity of RettBe 2.0 as well as for determining its clinical and functional significance. Finally, the investigators will obtain input from a panel of clinicians (site PIs and their designated clinicians) about content validity and clinical impact. The resulting version will be released as RettBe 3.0.

DETAILED DESCRIPTION:
Behavioral abnormalities, ranging from autistic symptoms to anxiety and mood lability, are now recognized as major clinical issues in RTT. These clinical manifestations are particularly problematic in higher functioning individuals since they seem to substantially affect their quality of life. Moreover, novel drug treatments aiming at RTT's neurobiological mechanisms have the potential of targeting these abnormal behaviors. Despite the recent emphasis on abnormal behaviors, little is known about their characteristics, severity, and impact. This is due, in part, to the paucity of behavioral measures compatible with the cognitive and motor impairments of RTT. The investigators currently have only one instrument with limited validation for delineating the range of behavioral abnormalities in RTT (the parent-rated Rett Syndrome Behavioral Questionnaire (RSBQ)), which is a significant shortcoming to the implementation of treatment trials. Moreover, there has not been a systematic approach for defining behavioral abnormalities in RTT (e.g., definition of mood abnormalities in RTT). These deficiencies have led the investigators to propose the creation of a broad-based behavioral outcome measure for use in RTT at different ages. Due to the complexity of the clinical evolution of RTT and the relative limited knowledge on its adult period, the investigators will focus on children with RTT ages 3-18 years. The new measure will allow for standardized quantifications of behavioral outcomes in treatment trials and, eventually, in clinical practice. The investigators recognize that developing an instrument with strong psychometric properties is a major endeavor; therefore, the investigators conceived this project as a multi-stage process.

The first stage, conducted with support of Rettsyndrome.org, consisted of developing a prototype or first version of a behavioral questionnaire for parents of children with RTT (3-18 years), which the investigators have termed RettBe 1.0. The initial part of this study will test the psychometric properties (i.e., structure, content validity) of RettBe 1.0 with an initial cohort of 100 participants. This stage intends to transform RettBe 1.0 into a fully developed behavioral instrument within the framework of the Natural History Study (RTT5211). Thus, in Aim 1 the investigators will evaluate psychometrically RettBe 1.0 following, in part, previous studies including their examination of anxiety instruments and adaptation of the Anxiety, Depression and Mood Scale (ADAMS) for RTT, and their adaptations of the Aberrant Behavior Checklist-Community (ABC-C) for fragile X syndrome and Down syndrome. In Aim 1, they will also refine RettBe 1.0 by adding new "missing" items based on parental input or clinician (PIs of sites involved) feedback. The resulting instrument, RettBe 2.0 will be tested in Aim 2.

Testing of RettBe 2.0 will be carried out with a new (naïve) validation cohort of 300 subjects and two raters (preferentially both parents/caregivers, alternatively one teacher or therapist), to determine inter-rater reliability. One rater, preferentially a parent, will be asked to also complete three other behavioral measures (RSBQ, ADAMS, ABC-C) for comparisons. Scores for RettBe 2.0 will be analyzed in terms of psychometric properties, as performed for RettBe 1.0. However, in addition to structure (construct validity) and content validity, the investigators will also examine convergent and discriminant validity by correlating domain RettBe 2.0 scores with those of comparable and non-comparable domain scores of the RSBQ, ADAMS, and ABC-C, respectively.

Finally, Aim 3 will use data from the RTT5211 protocol to determine the effect of age on RettBe 2.0 scores and the clinical and functional significance of the measure. Specifically, the investigators will examine score distributions throughout the age range, with special emphasis on early childhood (3-8 years), late childhood (8-12 years), and adolescence (>12 years). Clinical and functional relevance will be determined by correlations with instruments measuring multiple parameters of clinical severity, specifically, the CGI-S, Clinical Severity Scale, and Motor Behavior Assessment. Relevance to quality of life will be evaluated by correlations with the Child Health Questionnaire-Parent Form 50 (CHQ-PF50; child-oriented measure) and The Short Form (36) Health Survey (SF-36v2TM Health Survey; parent-oriented measure). All these instruments are components of the core RTT5211 protocol. Finally, prior to its release as RettBe 3.0 (if psychometric properties are good-excellent), the investigators will obtain input from a panel of clinicians (site PIs and their designated clinicians) about content validity and clinical impact.

ELIGIBILITY:
Inclusion Criteria

RettBe 1.0 Initial Cohort:

* Females 3 - 18 years
* Meets revised 2010 diagnostic criteria for classic or atypical RTT
* Post-regression status
* Documentation of positive MECP2 mutation
* Enrolled in the Natural History Study (RTT5211)

RettBe 2.0 Validation Cohort:

* Meet above criteria
* Two raters are available and willing to evaluate the subject
* Must not have participated in RettBe 1.0

Exclusion Criteria

Both RettBe 1.0 and RettBe 2.0:

* Do not meet the above inclusion criteria
* Foster children
* Non-English speakers

Ages: 3 Years to 18 Years | Sex: Female
Age Groups: Child, Adult
Study Population: A total of 400 subjects with RTT between the ages of 3 and 18 years of age will be recruited from RTT5211, which collects longitudinal clinical and neurobehavioral data in RTT and related disorders. This study will only include participants who meet 2010 diagnostic criteria for classic or atypical RTT and have a MECP2 mutation.
  Recruitment into this study will come from the larger cohort of those enrolled in the Natural History Study (RTT5211), a study aiming at enrolling 1000 participants with RTT. As a part of the Natural History Study (RTT5211), subjects provide their email address. RTT5211 participants will be emailed an invitation to join this study. Consent and study participation will be done online via a unique link in the invitation.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
RettBE 1.0 Score | 8 months
  Scores from RettBe 1.0, a 50-item questionnaire will be analyzed for psychometric properties, including content validity. RettBe 1.0 scores will be subjected to factor analysis to ensure domain-appropriate balance and structure.
RettBe 2.0 Score | 8 months
  RettBe 2.0 will be analyzed for psychometric properties. In addition, these raters will be completing other behavioral and clinical/functional measures for further evaluating the validity of RettBe 2.0 as well as for determining its clinical and functional significance (Aim 3). RettBe 2.0 will be subjected to factor analysis to ensure domain-appropriate balance and structure.
RettBe 3.0 Score | 8 months
  RettBe 3.0 scores will be subjected to factor analysis to ensure domain-appropriate balance and structure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neul JL, Kaufmann WE, Glaze DG, Christodoulou J, Clarke AJ, Bahi-Buisson N, Leonard H, Bailey ME, Schanen NC, Zappella M, Renieri A, Huppke P, Percy AK; RettSearch Consortium. Rett syndrome: revised diagnostic criteria and nomenclature. Ann Neurol. 2010 Dec;68(6):944-50. doi: 10.1002/ana.22124. PMID 21154482
- [Background] Robertson L, Hall SE, Jacoby P, Ellaway C, de Klerk N, Leonard H. The association between behavior and genotype in Rett syndrome using the Australian Rett Syndrome Database. Am J Med Genet B Neuropsychiatr Genet. 2006 Mar 5;141B(2):177-83. doi: 10.1002/ajmg.b.30270. PMID 16389588
- [Background] Lane JB, Lee HS, Smith LW, Cheng P, Percy AK, Glaze DG, Neul JL, Motil KJ, Barrish JO, Skinner SA, Annese F, McNair L, Graham J, Khwaja O, Barnes K, Krischer JP. Clinical severity and quality of life in children and adolescents with Rett syndrome. Neurology. 2011 Nov 15;77(20):1812-8. doi: 10.1212/WNL.0b013e3182377dd2. Epub 2011 Oct 19. PMID 22013176
- [Background] Cobb S, Guy J, Bird A. Reversibility of functional deficits in experimental models of Rett syndrome. Biochem Soc Trans. 2010 Apr;38(2):498-506. doi: 10.1042/BST0380498. PMID 20298210
- [Background] Kaufmann WE, Tierney E, Rohde CA, Suarez-Pedraza MC, Clarke MA, Salorio CF, Bibat G, Bukelis I, Naram D, Lanham DC, Naidu S. Social impairments in Rett syndrome: characteristics and relationship with clinical severity. J Intellect Disabil Res. 2012 Mar;56(3):233-47. doi: 10.1111/j.1365-2788.2011.01404.x. Epub 2011 Mar 8. PMID 21385260
- [Background] Aman MG, Singh NN (1986) Aberrant Behavior Checklist-Community manual. East Aurora, NY: Slosson Educational publications.
- [Background] Sansone SM, Widaman KF, Hall SS, Reiss AL, Lightbody A, Kaufmann WE, Berry-Kravis E, Lachiewicz A, Brown EC, Hessl D. Psychometric study of the Aberrant Behavior Checklist in Fragile X Syndrome and implications for targeted treatment. J Autism Dev Disord. 2012 Jul;42(7):1377-92. doi: 10.1007/s10803-011-1370-2. PMID 21972117
- [Background] Ji NY, Capone GT, Kaufmann WE. Autism spectrum disorder in Down syndrome: cluster analysis of Aberrant Behaviour Checklist data supports diagnosis. J Intellect Disabil Res. 2011 Nov;55(11):1064-77. doi: 10.1111/j.1365-2788.2011.01465.x. Epub 2011 Aug 30. PMID 21883598
- [Background] Barnes KV, Coughlin FR, O'Leary HM, Bruck N, Bazin GA, Beinecke EB, Walco AC, Cantwell NG, Kaufmann WE. Anxiety-like behavior in Rett syndrome: characteristics and assessment by anxiety scales. J Neurodev Disord. 2015;7(1):30. doi: 10.1186/s11689-015-9127-4. Epub 2015 Sep 15. PMID 26379794
- [Background] Mount RH, Charman T, Hastings RP, Reilly S, Cass H. The Rett Syndrome Behaviour Questionnaire (RSBQ): refining the behavioural phenotype of Rett syndrome. J Child Psychol Psychiatry. 2002 Nov;43(8):1099-110. doi: 10.1111/1469-7610.00236. PMID 12455930
- [Background] Mount RH, Hastings RP, Reilly S, Cass H, Charman T. Behaviour problems in adult women with Rett syndrome. J Intellect Disabil Res. 2002 Nov;46(Pt 8):619-24. doi: 10.1046/j.1365-2788.2002.00442.x. PMID 12427169
- [Background] Khwaja OS, Ho E, Barnes KV, O'Leary HM, Pereira LM, Finkelstein Y, Nelson CA 3rd, Vogel-Farley V, DeGregorio G, Holm IA, Khatwa U, Kapur K, Alexander ME, Finnegan DM, Cantwell NG, Walco AC, Rappaport L, Gregas M, Fichorova RN, Shannon MW, Sur M, Kaufmann WE. Safety, pharmacokinetics, and preliminary assessment of efficacy of mecasermin (recombinant human IGF-1) for the treatment of Rett syndrome. Proc Natl Acad Sci U S A. 2014 Mar 25;111(12):4596-601. doi: 10.1073/pnas.1311141111. Epub 2014 Mar 12. PMID 24623853
- [Background] Vignoli A, Fabio RA, La Briola F, Giannatiempo S, Antonietti A, Maggiolini S, Canevini MP. Correlations between neurophysiological, behavioral, and cognitive function in Rett syndrome. Epilepsy Behav. 2010 Apr;17(4):489-96. doi: 10.1016/j.yebeh.2010.01.024. Epub 2010 Mar 16. PMID 20236870
- [Background] Berry-Kravis E, Hessl D, Abbeduto L, Reiss AL, Beckel-Mitchener A, Urv TK; Outcome Measures Working Groups. Outcome measures for clinical trials in fragile X syndrome. J Dev Behav Pediatr. 2013 Sep;34(7):508-22. doi: 10.1097/DBP.0b013e31829d1f20. PMID 24042082
- [Background] Norris M, Lecavalier L. Evaluating the use of exploratory factor analysis in developmental disability psychological research. J Autism Dev Disord. 2010 Jan;40(1):8-20. doi: 10.1007/s10803-009-0816-2. Epub 2009 Jul 17. PMID 19609833